CLINICAL TRIAL: NCT04856085
Title: A Phase 2 Study to Evaluate the Safety, Tolerability, and Efficacy of Regimens Containing VIR-2218, VIR-3434, and/or PEG-IFNα in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: Study of VIR-2218, VIR-3434, and/or PEG-IFNα in Subjects With Chronic Hepatitis B Virus Infection
Acronym: MARCH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-2218-1006
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (13):
- Cohort 1a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple lead-in doses of VIR-2218, then combination therapy with VIR-2218 + VIR-3434 for 20 weeks total
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 2a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple lead-in doses of VIR-2218, then combination therapy with VIR-2218 + VIR-3434 for 20 weeks total
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 3a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for 4 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 4a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for 4 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 5a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for 11 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 6a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for 11 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 7a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for 44 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 8a (VIR-2218 + VIR-3434) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 for 20 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 1b (VIR-3434) (Experimental): Participants will receive multiple doses of VIR-3434 for 44 weeks
  Interventions: Drug: VIR-3434
- Cohort 2b (VIR-3434) (Experimental): Participants will receive multiple doses of VIR-3434 for 20 weeks
  Interventions: Drug: VIR-3434
- Cohort 1c (VIR-2218 + VIR-3434 + PEG-IFNα) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 + PEG-IFNα for 24 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434; Drug: PEG-IFNα
- Cohort 2c (VIR-2218 + VIR-3434 + PEG-IFNα) (Experimental): Participants will receive multiple doses of VIR-2218 + VIR-3434 + PEG-IFNα for 48 weeks
  Interventions: Drug: VIR-2218; Drug: VIR-3434; Drug: PEG-IFNα
- Cohort 1d (VIR-3434 + PEG-IFNα) (Experimental): Participants will receive multiple doses of VIR-3434 + PEG-IFNα for 48 weeks
  Interventions: Drug: VIR-3434; Drug: PEG-IFNα

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Other Names: Elebsiran
  Arms: Cohort 1a (VIR-2218 + VIR-3434); Cohort 1c (VIR-2218 + VIR-3434 + PEG-IFNα); Cohort 2a (VIR-2218 + VIR-3434); Cohort 2c (VIR-2218 + VIR-3434 + PEG-IFNα); Cohort 3a (VIR-2218 + VIR-3434); Cohort 4a (VIR-2218 + VIR-3434); Cohort 5a (VIR-2218 + VIR-3434); Cohort 6a (VIR-2218 + VIR-3434); Cohort 7a (VIR-2218 + VIR-3434); Cohort 8a (VIR-2218 + VIR-3434)
Drug: VIR-3434 — VIR-3434 given by subcutaneous injection
  Other Names: Tobevibart
Drug: PEG-IFNα — PEG-IFNα given by subcutaneous injection
  Arms: Cohort 1c (VIR-2218 + VIR-3434 + PEG-IFNα); Cohort 1d (VIR-3434 + PEG-IFNα); Cohort 2c (VIR-2218 + VIR-3434 + PEG-IFNα)

SUMMARY:
This is a phase 2 study in which participants with chronic hepatitis B virus (HBV) infection will receive VIR-2218, VIR-3434 and/or PEG-IFNα and be assessed for safety, tolerability, and efficacy

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 - <66 years
* Chronic HBV infection for >/= 6 months
* On NRTI therapy for >/= 2 months at the time of screening

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the participant unsuitable for participation
* Significant fibrosis or cirrhosis
* History or evidence of drug or alcohol abuse
* History of chronic liver disease from any cause other than chronic HBV infection
* History of hepatic decompensation
* History of anaphylaxis
* History of allergic reactions, hypersensitivity, or intolerance to monoclonal antibodies, antibody fragments, or any excipients of VIR-3434
* History of immune complex disease
* History of known contraindication to any interferon product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (TEAEs) | Up to 72 weeks
Proportion of participants with serious adverse events (SAEs) | Up to 72 weeks
Proportion of participants with hepatitis B surface antigen (HBsAg) loss (defined as undetectable HBsAg) at end of treatment | Up to 48 weeks
Proportion of participants with HBsAg loss (defined as undetectable HBsAg) at 24 weeks post-end of treatment | Up to 72 weeks

SECONDARY OUTCOMES:
Absolute serum HBsAg and change from baseline across all timepoints in the study | Up to 110 weeks
Nadir and maximum reduction of serum HBsAg from baseline | Up to 110 weeks
Proportion of participants achieving sustained suppression of HBV DNA (< lower limit of quantification (LLOQ) for >= 24 weeks after discontinuation of all treatment, including NRTIs) | Up to 110 weeks
For hepatitis B e-antigen (HBeAg)-positive participants: Proportion of participants with HBeAg loss (undetectable HBeAg) and/or anti-HBe seroconversion at any timepoint | Up to 110 weeks
For HBeAg-positive participants: Time to HBeAg loss (undetectable HBeAg) and/or anti-HBe seroconversion | Up to 110 weeks
Cmax | Up to 110 weeks
AUClast | Up to 110 weeks
t1/2 | Up to 110 weeks
CL/F | Up to 110 weeks
Number of participants with incidence and titers of anti-drug antibody (ADA) (if applicable) to VIR-3434 | Up to 110 weeks
Proportion of participants meeting criteria for nucleotide reverse transcriptase inhibitors (NRTI) discontinuation | Up to 60 weeks
Proportion of participants meeting criteria for NRTI retreatment | Up to 110 weeks
Proportion of participants achieving undetectable HBsAg and sustained suppression of HBV DNA [below the LLOQ, target not detected (TND)] >/= 24 weeks after discontinuation of all treatment, including NRTIs | Up to 110 weeks
Proportion of participants with serum HBsAg < 10 IU/mL at end of treatment | Up to 48 weeks
Proportion of participants with serum HBsAg < 10 IU/mL at 24 weeks post-end of treatment | Up to 72 weeks
  48 weeks treatment + 24 weeks post-end of treatment
Proportion of participants with anti-HBs seroconversion | Up to 110 weeks
Time to achieve nadir of serum HBsAg | Up to 110 weeks
Time to achieve serum HBsAg loss | Up to 110 weeks

CONTACTS AND LOCATIONS:
Locations (32):
- United States (5):
  - Investigative Site, San Francisco, California
  - Investigative Site, Miami, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Hillsborough, New Jersey
- Canada (2):
  - Investigative Site, Toronto
  - Investigative Site, Vancouver
- Germany (3):
  - Investigative Site, Frankfurt
  - Investigative Site, Hanover
  - Investigative Site, Mannheim
- Hong Kong (3):
  - Investigative Site, Hong Kong, Shatin
  - Investigative Site, Hong Kong, Tai Po District
  - Investigative Site, Hong Kong
- Investigative Site, Kuala Lumpur, Malaysia
- Investigative Site, Chisinau, Moldova
- New Zealand (4):
  - Investigative Site, Auckland
  - Investigative Site, Hamilton
  - Investigative Site, Tauranga
  - Investigative Site, Wellington
- Investigative Site, Bucharest, Romania
- South Korea (3):
  - Investigative Site, Busan
  - Investigative Site, Seoul
  - Investigative Site, Yangsan
- Taiwan (5):
  - Investigative Site, Chiayi City
  - Investigative Site, Kaohsiung City
  - Investigative Site, Taichung
  - Investigative Site, Taipei
  - Investigative Site, Taoyuan
- Investigative Site, Kyiv, Ukraine
- United Kingdom (3):
  - Investigative Site, Birmingham
  - Investigative Site, London
  - Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No